CLINICAL TRIAL: NCT05557383
Title: Department of Nursing Hui-Chin Chen Head Nurse
Brief Title: Effect of Using Peanut Ball on the Length of Labor for Women Laboring With an Epidural
Acronym: peanutball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CG19310B
Record Dates: First submitted 2022-09-13; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2019-10

CONDITIONS: Labor; Epidural Anesthesia
Keywords: peanut ball; Length of Labor

STUDY DESIGN:
Intervention Model Description: A two-group controlled, randomized study, the intervention groups: use peanut ball, control groups: not use peanut ball
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes Assessor has no information for use peanut ball
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use peanut ball (Experimental): Registered nurses were educated by the investigators on the study protocol, and standard care was given to both the intervention and control groups.The peanut ball was placed between the legs of a woman in the intervention group immediately after she received her epidural and consented to participate in the study.
  Interventions: Behavioral: use peanut ball
- usual care (No Intervention): usual nursing care.

INTERVENTIONS:
Behavioral: use peanut ball — The peanut ball was placed between the legs of a woman in the intervention group immediately after she received her epidural and consented to participate in the study.
  Other Names: usual care
  Arms: use peanut ball

SUMMARY:
The purpose of this study is to investigate the Effect of using peanut ball on the length of labor, delivery pattern and childbirth satisfaction for women laboring with an Epidural.This study aims to understand the intervention of using peanut ball in the future during the delivery period is expected.it is expected to reduce the cesarean section with delayed delivery.

DETAILED DESCRIPTION:
In this study, expectant mothers who used epidural anesthesia to reduce pain during delivery in the delivery room of a central medical center, including primiparous women and menstrual women, were evaluated for compliance with the acceptance criteria through the mother's manual and maternity examination data. The maternal agreed to fill out the subject consent form,After obtaining the consent form of the test subject, it is included in the research object of this trial. It is expected that 190 expectant mothers will be accepted, and 40 expectant mothers will be accepted. The research tool uses the Chinese version of the Mackey Childbirth Satisfaction Rating Scale to measure women's satisfaction with the behavioral performance of self, partner, and baby during delivery / production. The scale was agreed by the original author and translator. Use consists of six levels: overall satisfaction (3 questions), self-satisfaction (9 questions), newborns (3 questions), midwifery care workers (9 questions), physicians (6 questions), and Satisfaction with partners (2 questions), a total of 32 items. After data collection, the data will be archived and analyzed with Statistical Package for the Social Sciences (version 22.0) software.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 20 years old
2. Full-term women who are more than 37 weeks pregnant and diagnosed as low-risk pregnancy by physicians
3. Pain relief with epidural anesthesia
4. Singleton
5. Normal birth position ( The first part of the head)
6. Know the Chinese characters and be able to communicate in Chinese and Taiwanese
7. Agree to participate in this researcher.

Exclusion Criteria:

1. Language communication barriers
2. Any abnormality and comorbidity of the woman and fetus during labor
3. No epidural anesthesia for pain relief.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Laboring women were recruited if they met the inclusion criteria, which included being in active labor, using an epidural for pain control
Enrollment: 190 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Correlation between peanut ball intervention and labor progress | Record the time of the first and second stage of labor.Data collect through study completion about 1 year. analysis with SPSS.Because the data were tested for non-normal distribution, Mann-Whitney U test (continuous variable) and χ2 (discontinuous variab
  If assign to the experimental group, will provide peanut ball interventions every 30 minutes, and assist in changing postures according to the mother's wishes, including four position. Each time the peanut balls are placed for at least 10 minutes, continuous electronic fetal monitoring is given, and the uterine contractions and fetal conditions of the expecting mother are assessed every 30 minutes. When the cervix full dilates, and fetal descends, stop using the peanut balls and be ready to labor. Control group: no intervention with peanut balls, regular care as experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No